CLINICAL TRIAL: NCT03645551
Title: Clinical Longevity of Ceramic Laminate Veneers Bonded to Teeth With and Without Existing Composite Restorations up to 10 Years
Brief Title: Clinical Longevity of Ceramic Laminate Veneers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Marco Gresnigt, independent investigator, University Medical Center Groningen
Other Study IDs: Gresnigt
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: dentistry; laminate veneer; existing restoration; survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: checkup, no test — In this study we would like to examine if existing restorations already applied in teeth which we treated with laminate veneers had an effect. We will evaluate the laminate veneers by sight and take pictures and use a questionnaire

SUMMARY:
Rationale: Survival rates of teeth with laminate veneers were reported to have more marginal caries and discoloration when existing restorations are present. However in these studies no conditioning of the existing restorations was performed.

Objective: This study evaluate the survival rate of ceramic laminate veneers bonded to teeth with and without existing composite restorations Study design: Prospectief Cohort research Study population: the participants received laminate veneers and older then 18 years.

Intervention (if applicable): The participants received laminate veneers in the past. No intervention.

Main study parameters/endpoints: Survival and success of laminate veneers with existing restorations: Survival (no loss of laminate veneer during follow up time), Success was measured using USPHS health criteria.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The participants are asked to come for a check-up of their restorations, the investigators will evaluate the laminate veneers by sight and take some light photo's and a patient questionnaire will be given.

DETAILED DESCRIPTION:
The use of ceramic laminate veneers as opposed to metal-ceramic or all-ceramic full-coverage crowns is a minimal invasive treatment option in reconstructive dentistry. Since their retention relies solely on adhesion, durable adhesion of resin luting cements to both the enamel/dentin and the cementation surface of the ceramic is crucial. Luting cements used in conjunction with phosphoric acid etching followed by adhesive application on enamel show reliable adhesion with mean bond strengths up to 40 MPa. Also, etching the intaglio of glass ceramic veneers with hydrofluoric acid followed by silane coupling agent application delivers bond strength values similar to or higher than to enamel. Even after long-term water storage and thermocycling aging conditions, promising results were reported with resin-ceramic adhesion. Ceramic laminates are indicated not only to restore malformed, malpositioned, or discolored teeth where mainly the substrate is the enamel and/or dentin but also in situations where resin composite restorations are present on the tooth to be restored. In case of secondary caries, severe marginal or surface changes, it may be necessary to remove such restorations. On the other hand, degradation of polymers in the aggressive oral environment may decrease the free radicals available on the resin surface that may eventually decrease the adhesion of resin cements to such composites. However, limited information is available on the survival of ceramic laminates on such existing composite restorations where mainly fractures and marginal defects were reported. Defects were especially noticed at the locations where the existing fillings were present. In fact, today, advances in surface conditioning methods and adhesion promoters enable durable composite-composite adhesion. Among numerous other methods, several studies reported increased composite- composite bond strengths after conditioning the composites with alumina or alumina-coated silica particles followed by silanization. The process of silanization promotes the wettability of the substrates and further reacts with the glass particles present on the composite surface forming covalent bonds. Composite- composite bond strength simulating aging after silica coating and silanization was reported to deliver significantly higher bond strengths (46-52 MPa) than conditioning the composite substrate with phosphoric acid and adhesive resin application only (16-25 MPa). Unfortunately, the previous clinical studies did not report application of any surface conditioning method prior to cementation of ceramic laminates. In clinical practice, the clinical dilemma is whether or not to remove the existing composite restorations with no indications of caries or acceptable surface degradation that could be refinished and repolished. Alternatively, full-coverage crowns are indicated on teeth with large composite restorations that require more tissue removal yielding to preparations in dentin that is a substrate less favorable to bond onto than enamel. The objective of this prospective clinical study is to evaluate the performance of ceramic laminate veneers bonded onto either intact teeth or to teeth with existing composite restorations with no indications of caries, ditching, or marginal staining. The null hypothesis tested is that the presence of existing composite restorations would not decrease the survival rate of ceramic laminate veneers compared to those bonded onto intact teeth.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with laminate veneers by dr. Gresnigt
* at least 18 years old
* able to read and sign the informed consent document
* physically and psychologically able come for an evaluation as outlined by the investigators.

Exclusion Criteria:

* People not able to return or not willing to come for an evaluation
* People died

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an evaluative prospective study where over 450 laminate veneers were made in 110 patients. All patients will be asked to enrol in the study. Probably 90% will come to an evaluation appointment when asked to enrol. 90% seems very high but all patients were formerly patients when dr. Gresnigt was still working in a private general dentistry office. So reasonably 400 laminate veneers with 100 patients will be expected to be evaluated.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Restorations which survived when applied on the tooth till the last follow up. (survival) | june 2007- september 2018
  Caries, debonding, chipping, and fracture are considered as absolute failures. Due to these factors the restorations will be lost and a new one has to be made, that is why these scores are survival and main endpoints.

SECONDARY OUTCOMES:
Succes | june 2007 - september 2018
  Both observers evaluate the restorations independently, according to the modified United States Public Health Service (USPHS) criteria on Marginal Adaptation, Color match, Marginal discoloration, Surface roughness, Fracture of the restoration, Fracture of the tooth, wear of the restoration, wear of the antagonist, Caries, Postoperative sensitivity. Patient satisfaction. Above scores are not indications for removal of the restoration but sometimes can be a deterioration of the restoration itself. So the esthetic outcome can be a little less but the survival is still good.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Cune, Prof, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: No
This study will focus on laminate veneers bonded to teeth with and without composite restorations. And also will be looked at preparations were more than 50% of dentin was exposed if an immediate dentin sealing would have an benefit.

REFERENCES:
- [Background] Peumans M, De Munck J, Fieuws S, Lambrechts P, Vanherle G, Van Meerbeek B. A prospective ten-year clinical trial of porcelain veneers. J Adhes Dent. 2004 Spring;6(1):65-76. PMID 15119590
- [Background] Gresnigt MMM, Ozcan M, Carvalho M, Lazari P, Cune MS, Razavi P, Magne P. Effect of luting agent on the load to failure and accelerated-fatigue resistance of lithium disilicate laminate veneers. Dent Mater. 2017 Dec;33(12):1392-1401. doi: 10.1016/j.dental.2017.09.010. Epub 2017 Nov 1. PMID 29079354
- [Background] Gresnigt MM, Cune MS, de Roos JG, Ozcan M. Effect of immediate and delayed dentin sealing on the fracture strength, failure type and Weilbull characteristics of lithiumdisilicate laminate veneers. Dent Mater. 2016 Apr;32(4):e73-81. doi: 10.1016/j.dental.2016.01.001. Epub 2016 Feb 5. PMID 26856454
- [Background] Gresnigt MM, Kalk W, Ozcan M. Randomized clinical trial of indirect resin composite and ceramic veneers: up to 3-year follow-up. J Adhes Dent. 2013 Apr;15(2):181-90. doi: 10.3290/j.jad.a28883. PMID 23534025
- [Background] Gresnigt MM, Kalk W, Ozcan M. Clinical longevity of ceramic laminate veneers bonded to teeth with and without existing composite restorations up to 40 months. Clin Oral Investig. 2013 Apr;17(3):823-32. doi: 10.1007/s00784-012-0790-5. Epub 2012 Jul 21. PMID 22821429
- [Background] Gresnigt M, Ozcan M, Kalk W. Esthetic rehabilitation of worn anterior teeth with thin porcelain laminate veneers. Eur J Esthet Dent. 2011 Autumn;6(3):298-313. PMID 21876866
- [Background] Gresnigt MM, Ozcan M, Kalk W, Galhano G. Effect of static and cyclic loading on ceramic laminate veneers adhered to teeth with and without aged composite restorations. J Adhes Dent. 2011 Dec;13(6):569-77. doi: 10.3290/j.jad.a21742. PMID 21734979
- [Derived] Gresnigt MMM, Cune MS, Schuitemaker J, van der Made SAM, Meisberger EW, Magne P, Ozcan M. Performance of ceramic laminate veneers with immediate dentine sealing: An 11 year prospective clinical trial. Dent Mater. 2019 Jul;35(7):1042-1052. doi: 10.1016/j.dental.2019.04.008. Epub 2019 May 10. PMID 31084936